CLINICAL TRIAL: NCT07194304
Title: Effect of Parenteral Alpha-Tocopherol in the Definitive Surgery of Tetralogy of Fallot
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Suprayitno Wardoyo, Consultant Cardiothoracic Surgeon, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET-273/UN2.F1/ETIK/PPM.00.02/
Record Dates: First submitted 2025-07-04; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Tetralogy of Fallot (TOF); Alpha-tocopherol; Cardiac Surgery
Keywords: TOF; alpha-tocopherol; cardiac surgery; troponin I
MeSH Terms: conditions — Tetralogy of Fallot | interventions — alpha-Tocopherol; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- alpha-tocopherol (Experimental): assigned to receive either parenteral alpha-tocopherol (4 mg/kg)
  Interventions: Drug: alpha-Tocopherol
- sterile water for injection (Placebo Comparator): the control group received a placebo (sterile water for injection/aquabidest)
  Interventions: Drug: Sterile Water for Injection

INTERVENTIONS:
Drug: alpha-Tocopherol — patients in the intervention group received parenteral alpha-tocopherol at a dose of 4 mg/kg body weight
  Arms: alpha-tocopherol
Drug: Sterile Water for Injection — the control group received a placebo (sterile water for injection/aquabidest)
  Arms: sterile water for injection

SUMMARY:
Introduction:

Tetralogy of Fallot (ToF) correction with cardiopulmonary bypass (CPB) poses a risk of ischemia-reperfusion injury, especially in cyanotic myocardium. Alpha-tocopherol, a potent antioxidant, may reduce myocardial damage during surgery.

Methods:

This randomized controlled trial included 58 ToF patients aged 1-10 years undergoing definitive surgery with CPB at Integrated Heart Center, Cipto Mangunkusumo Hospital. Patients were randomly assigned to receive either parenteral alpha-tocopherol (4 mg/kg) or placebo at the initiation of CPB. The primary outcome was postoperative troponin I level.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital heart disease Tetralogy of Fallot (ToF)
* Age between 1 and 10 years
* Scheduled for definitive repair of ToF using cardiopulmonary bypass (CPB) at PJT-RSCM

Exclusion Criteria:

* History of prior palliative surgery (e.g., Blalock-Taussig shunt)
* Presence of additional congenital heart disease requiring major modification or addition of surgical procedures
* History of central nervous system disorder or stroke
* History of cardiopulmonary resuscitation (CPR)
* Undergoing redo surgery (e.g., residual stenosis, bleeding)

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Serum Troponin I Concentration (ng/L) | Before surgery, 1 hour after surgery, and 8 hours after surgery
  Serum Troponin I concentration will be measured at baseline (before surgery), 1 hour after surgery, and 8 hours after surgery to assess the extent of myocardial injury associated with cardiopulmonary bypass during Tetralogy of Fallot repair.

SECONDARY OUTCOMES:
Change in Serum Malondialdehyde (MDA) Concentration (ng/mL) | Before surgery, 1 hour after surgery, and 8 hours after surgery
  Serum malondialdehyde (MDA), a biomarker of oxidative stress, will be measured at baseline (before surgery), 1 hour after surgery, and 8 hours after surgery to evaluate oxidative injury associated with cardiopulmonary bypass during Tetralogy of Fallot repair.
Change in Serum Lactate Concentration (mmol/L) | Before surgery, 1 hour, 6 hours, 12 hours, and 24 hours after surgery
  Serum lactate levels will be measured at baseline (before surgery), and at 1 hour, 6 hours, 12 hours, and 24 hours after surgery to evaluate tissue perfusion and metabolic response associated with cardiopulmonary bypass during Tetralogy of Fallot repair.
Myocardial Injury Score (Histopathology, Scale 0-3) | 15 minutes after release of the aortic cross-clamp
  Myocardial tissue injury will be assessed from biopsy samples collected 15 minutes after release of the aortic cross-clamp. Injury will be graded on a histopathological scale ranging from 0 to 3, where 0 = no injury and 3 = severe injury. Higher scores indicate worse myocardial damage.
Apoptotic Index (% of Apoptotic Cardiomyocytes) | tissue sample is collected 15 minutes after releasing the aortic cross clamp
  The apoptotic index will be calculated from myocardial tissue samples collected 15 minutes after release of the aortic cross-clamp. Sections are stained with TUNEL and examined at 40× magnification across 6 hotspot areas. The index is expressed as the percentage of TUNEL-positive cardiomyocytes per 100 cardiomyocytes. The scale ranges from 0% (no apoptosis) to 100% (all cells apoptotic). Higher values indicate greater myocardial apoptosis.
Duration of Mechanical Ventilation (hours) | From end of surgery until extubation
  Duration of postoperative mechanical ventilation will be recorded in hours.
anti-cTnI | tissue sample is collected 15 minutes after releasing the aortic cross clamp
GPx expression | tissue sample is collected 15 minutes after releasing the aortic cross clamp
Intensive Care Unit Length of Stay (days) | From ICU admission until ICU discharge, assessed up to 14 days
  ICU length of stay will be recorded in days from ICU admission until ICU discharge.
Hospital Length of Stay (days) | From hospital admission until hospital discharge, assessed up to 30 days
  Hospital length of stay will be recorded in days from hospital admission until discharge.
Vasoactive-Inotropic Score (VIS, Scale 0-X) | First 24 hours after surgery
  Vasoactive-Inotropic Score (VIS) will be calculated to quantify the amount of vasoactive support required after surgery. The VIS scale ranges from 0 to an open-ended maximum value; higher scores indicate greater need for vasoactive support and worse hemodynamic status.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No